CLINICAL TRIAL: NCT03060850
Title: A Phase I Study of AC0010 in Patients With Relapsed or Refractory CLL/SLL, MCL, DLBCL and Other Non-Hodgkin B-Cell Lymphoma
Brief Title: A Phase I Study of AC0010 in Patients With CLL/ SLL, MCL, DLBCL and Other NHL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou ACEA Pharmaceutical Research Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC201602AVTN05
Record Dates: First submitted 2017-02-10; First posted 2017-02-23 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — abivertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AC0010MA (Experimental): This is dose escalation study. Patients will receive AC0010MA 200mg bid,300mg bid,400mg bid or 500mg bid by mouth (the dose escalation whether ended depends on DLT and occupancy) everyday until intolerable toxicity or disease progression
  Interventions: Drug: AC0010MA

INTERVENTIONS:
Drug: AC0010MA — Participants in the dose escalation cohorts will be treated with AC0010MA every 28 days
  Other Names: AC0010

SUMMARY:
This is an open label, dose escalation, phase I study to determine the recommended Phase 2 dose (PR2D) by assessing the DLT, safety and efficacy of AC0010 in patients with B-cell lymphoma.

DETAILED DESCRIPTION:
This is an open label, dose escalation, phase I study to determine the PR2D by assessing the DLT, safety and efficacy of AC0010 in patients with B-cell lymphoma. This study includes two parts. During Part 1 Dose Escalation, the "3+3" design will be applied. Dose escalation will begin at dose level 1 = 400 mg. This dose escalation will be followed by an exploratory expansion phase in 3 or 4 groups of 15~41 patients each (CLL group, MCL group, non-germinal center B cell-like DLBCL group, and/or FL/WM(macroglobulinemia) group). The study will further evaluate the safety and efficacy of AC0010 in these patients in each group

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 years and 75 years (included), and patients is over 60 years cannot have more than 3 kinds of heart, lung, liver and kidney complications
* Histological confirmed CLL/SLL, MCL, non-GCB DLBCL
* Measurable disease (NHL: At least 1 measurable site of disease [>1.5 centimeter [cm] in the long axis regardless of short axis measurement or >1.0 cm in the short axis regardless of long axis measurement, and clearly measurable in 2 perpendicular dimensions])
* In dose escalation phase, other NHL (FL、WM、MZL、BL) patients who are relapsed refractory disease after at least 1 line of previous systemic therapy could be enrolled
* Could supply stored For Formalin Fixed and Paraffin-Embedded (FFPE) slides or block to the lab for testing or could accept biopsy in the screening.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 2
* Any of the following hematology values within 14 days prior to inclusion and prior to the first dose of study drug :
* Absolute neutrophil count (ANC) >= 750 cells/µL(0.75 x 109/L) without growth factors within 7 days prior to the first dose of study drug
* Spontaneous Platelets count > 50,000 cells/mm3, exclude transfusion dependent thrombocytopenia
* Adequate heart, liver, lung and renal function:
* Alkaline phosphatase (ALP) <5* ULN
* Creatinine determined by serum creatinine levels <=1.5 * ULN or a calculated creatinine clearance of >= 50 mL/min
* LVEF≥50% as determined by Ultrasonic Cardiogram (UCG)
* Any prior treatment (chemotherapy, radiotherapy or ) must be completed over 30 days or 5 *half life from the screening; all toxicities related to prior anticancer therapies must be recovered to grade ≤ 1 (CTCAE v 4.03)
* Patients without central nervous system involvement
* Life expectancy of more than 6 months
* Women of childbearing potential must have a negative serum beta human chorionic gonadotropin (β-hCG) or urine pregnancy test negative at Screening
* Women without pregnant or breastfeeding

Exclusion Criteria:

* Past history of major surgery within 4 weeks before signing the Informed consent form (ICF)
* Patents with Central nervous system (CNS) lymphoma
* Patients with prolymphocytic leukemia, patients with Richter's syndrome or suspected with Richter's syndrome
* Known with primary mediastinal lymphoma • Previous treated with tyrosine kinase inhibitors (TKIs) (including BTK inhibitor) or within 3 months received mono-antibody treatment prior to the first dose of study drug
* Prior history of malignancies other than lymphoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the patient has been free of the disease for ≥ 3 years
* Use of any standard or experimental anti-cancer drug therapy within 30 days prior to the first dose of study drug
* Autotransplantation within 6 months prior to the first dose of study drug
* Known received allogeneic stem cell transplantation
* History of stroke or intracranial hemorrhage within 6 months prior to the first dose of study drug
* Requires treatment with anticoagulation with warfarin or equivalent vitamin K antagonists
* Condition that requires treatment with a strong cytochrome P450 3A4/5 (CYP3A4/5) inhibitor
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months prior to the first dose of study drug, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
* ECG showed abnormal PR, QT and QRS interval (defined as: 12 lead electrocardiogram QT interval corrected Bazett (QTcB) > 430 ms (male) or 450 ms (female), PR> 240 ms, QRS> 110 ms), and electrocardiogram in rhythm, conduction and morphology appeared on the clinical significance of abnormal, such as complete left bundle branch block, myocardial infarction occurred within 6 months; risk factors cause QTc prolongation such as heart failure, arrhythmia, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or first-degree relatives had less than 40 years of history of sudden death or bradycardia (heart rate less than 50 beats per minute)
* Known HIV, active Hepatitis C Virus (HCV; RNA polymerase chain reaction (PCR)-positive) or active Hepatitis B Virus infection (HBs Ag positive or DNA PCR-positive) or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics
* All toxicities related to prior anticancer therapies recovered to grade ≤ 1 (exclude any grade alopecia)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times upper limit of normal (ULN) and total bilirubin >1.5xULN
* Blood urea nitrogen (BUN) or Cr >1.5x upper limits of normal (ULN)
* Uncontrolled pericardial effusion and pleural effusion
* History of Parkinson's disease; cerebellar disorders or other motor related diseases; patients with a history of pancreatitis
* Investigator judgment that patient is unsuitable to participate in study
* Uncontrolled pleural and pericardial effusion.
* Pregnant and lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2017-03-17 (Actual); Primary Completion 2019-12-14 (Estimated); Study Completion 2020-12-14 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose | On cycle one, up to 28 days
  Determine the recommended phase II dose (RP2D) of AC0010 in patients with relapsed or refractory CLL/SLL, MCL, DLBCL and other Non-Hodgkin B-Cell lymphoma

SECONDARY OUTCOMES:
24 hours occupancy of AC0010 | 24 hours
  AC0010 occupancy of the Bruton's tyrosine kinase (BTK) active site up to 24 hours
Tolerability as measured by adverse events using CTCAE and clinical laboratory parameters | Approximately 36 months
  Evaluation of tolerability of AC0010 measured by number, nature and severity of Adverse Events using CTCAE Version 4.03
Tolerability as measured by number of subjects with dose limiting toxicities | on cycle one, up to 28 days
  Evaluation of tolerability of AC0010 measured by number of subjects with dose limiting toxicities (DLTs)treatment
Maximum tolerated dose (MTD) | on cycle one, up to 28 days
  Maximum Tolerated Dose (MTD) as measured by the number of dose-limiting toxicities in each dose level
Occupancy of AC0010 after continued treatment | On first 4 cycles，up to 4 months
  AC0010 occupancy of the BTK active site after continued treatment
Objective Response Rate (ORR) | Approximately 36 months
  Safety and efficacy data will take place at the analysis time point
Cmax | Day 1, Day 28, D112
  Determine peak plasma concentration (Cmax) after oral administration of AC0010
Tmax | 5 min before-dose and 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 1, 5 min before-dose and 2, 4, 8, 12 hours post-dose on Day 28, 5 min before-dose on Day 112
  Time to reach maximum observed plasma concentration
t1/2 | 5 min before-dose and 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 1, 5 min before-dose and 2, 4, 8, 12 hours post-dose on Day 28, 5 min before-dose on Day 112
  plasma decay half-life
AUC(0-t) | 5 min before-dose and 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 1, 5 min before-dose and 2, 4, 8, 12 hours post-dose on Day 28, 5 min before-dose on Day 112
  Area under the curve from time zero to the last quantifiable concentration
AUC(0-∞) | 5 min before-dose and 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 1, 5 min before-dose and 2, 4, 8, 12 hours post-dose on Day 28, 5 min before-dose on Day 112
  Area under the curve from time zero to extrapolated infinity

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, MD, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital,Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No